CLINICAL TRIAL: NCT05475665
Title: A Randomized, Double-blind, Multicenter, Placebo-control, Parallel Group Phase # Study to Evaluate the Efficacy and Safety of Irbesartan and Amlodipine Combined Therapy in Essential Hypertension Patients
Brief Title: Clinical Efficacy and Safety Evaluation of Irbesartan High and Amlodipine Combined Therapy in Essential Hypertension Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HD-AI-302
Record Dates: First submitted 2022-07-24; First posted 2022-07-27 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — Irbesartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irbesartan/Amlodipine (Experimental)
  Interventions: Drug: Irbesartan/Amlodipine
- Irbesartan (Active Comparator)
  Interventions: Drug: Irbesartan

INTERVENTIONS:
Drug: Irbesartan/Amlodipine — Irbesartan/Amlodipine once daily for 8 weeks
  Arms: Irbesartan/Amlodipine
Drug: Irbesartan — Irbesartan once daily for 8 weeks
  Arms: Irbesartan

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of Irbesartan and Amlodipine combined therapy in patients with essential hypertension inadequately controlled on Irbesartan monotherapy

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 19 years or older on screening
* Signed informed consent
* Patients with Essential Hypertension
* Other inclusion applied

Exclusion Criteria:

* Orthostatic hypotension with symptom
* Other exclusion applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2022-07-14 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-06-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mean sitting systolic blood pressure (mmHg) | Week 8

SECONDARY OUTCOMES:
Change form baseline in mean sitting systolic blood pressure (mmHg) | Week 4
Change form baseline in mean sitting diastolic blood pressure (mmHg) | Week 4, 8
Responder rate | Week 4, 8
Target blood pressure reach rate | Week 4, 8

CONTACTS AND LOCATIONS:
Locations (1):
- Hanyang University Seoul Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Lee HY, Min KW, Han KA, Kim JS, Ahn JC, Kim MH, Lee JB, Shin SH, Kim CJ, Kim KH, Cho DK, Choi J, Rhee MY, Her SH, Kim W, Na JO, Cho GY, Kim SY, Park GM, Lee BK, Jo SH, Lee BW, Sohn IS, Kim DI, Ihm SH, Lee SH, Chung JW, Cho EJ, Son JW, Oh SJ, Hwang JY, Jeong JO, Han KR, Yoon HJ, Seo SM, Chung WJ, Bae JW, Choi JH, Hyun BJ, Cha JE, Yoo SJ, Shin J. The Efficacy and Tolerability of Irbesartan/Amlodipine Combination Therapy in Patients With Essential Hypertension Whose Blood Pressure Were not Controlled by Irbesartan Monotherapy. Clin Ther. 2024 Jun;46(6):481-489. doi: 10.1016/j.clinthera.2024.04.004. Epub 2024 May 3. PMID 38704294